CLINICAL TRIAL: NCT07185152
Title: The Effect of Mechanical Vibration and Flick Tapping Methods in Reducing Pain During Hepatitis B Vaccine Administration in Infants
Brief Title: The Effect of Mechanical Vibration and Flick Tapping Methods in Reducing Pain in Infant Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berrin GOGER (Other)
Responsible Party: Sponsor-Investigator, Berrin GOGER, Lecturer, Gümüşhane Universıty
Organization: Gümüşhane Universıty (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-95674917-108.99-245388; TDK-2024-15853 (Other Grant/Funding Number: KTU RECTORATE (SRP Coordination Unit))
Record Dates: First submitted 2025-09-03; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Health Knowledge, Attitudes, Practice; Health Behavior
Keywords: Infant, Pain, Pediatric nursing, Vaccines, Vibration
MeSH Terms: conditions — Behavior; Health Behavior; Pain

STUDY DESIGN:
Intervention Model Description: There are 3 groups in the randomized controlled experimental study. Mechanical vibration method was applied to one group, flick tapping method was applied to one group, and one group was included in the study as a control group without any intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical Vibration group (Experimental): Babies randomized to the Mechanical Vibration group were subjected to vibration approximately 1 cm above the injection site with a mechanical vibration device before and during the vaccination procedure.
  Interventions: Other: mechanical vibration
- Flick tapping group (Experimental): Before the vaccination procedure, the vaccination site was placed on the nail of the middle finger in the babies randomized to the flick tapping group, and then the vaccination was stimulated with a quick tap using the upper nail part of the middle finger.
  Interventions: Other: Flick tapping
- Control groups (No Intervention): The routine vaccination procedure was administered to the infants in this group.

INTERVENTIONS:
Other: mechanical vibration — Mechanical vibration was applied to babies randomized to the mechanical vibration group before and during the vaccination procedure.
  Arms: Mechanical Vibration group
Other: Flick tapping — Before the vaccination procedure, the vaccination site was placed on the nail of the middle finger in the babies randomized to the flick tapping group, and then the vaccination was stimulated with a quick tap using the upper nail part of the middle finger.
  Arms: Flick tapping group

SUMMARY:
A research protocol examining the effect of vibration on the crying duration variable in needle-related medical procedures in newborns also predicted that vibration therapy would be effective in reducing pain caused by vaccine injection and shortening the newborn's crying time.

Flicking the injection site can be used to control pain in childhood. To date, only one experimental study testing the flick method has reported that the flick method applied before intramuscular injection had lower pain scores in babies during and after vaccination.

Studies show that the positive effects of both methods are mentioned. However, no study has been found to examine the effects of both methods on injection pain that may occur when the second dose of Hepatitis B vaccine is administered in the neonatal period and compare their effects. The fact that the effects of mechanical vibration and flicking methods as pain relief strategies on reducing pain, physiological parameters and crying duration have not been examined in this population before shows the deficiency in the literature.This study aimed to examine the effect of flicking the injection site before the second dose of the Hepatitis B vaccine applied to the anterior surface of the vastus lateralis muscle in infancy and applying mechanical vibration to the injection site throughout the vaccination procedure on acute pain, crying duration and physiological parameters that may occur due to intramuscular injection.

DETAILED DESCRIPTION:
Most tactile stimuli, such as vibration, have the potential to reduce pain because many large fibers are present in the skin. It is stated that mechanical vibration works primarily by turning off the ascending transmission of the nociceptive afferent nerve signal in the spinal-thalamic pathway and may provide an alternative or additional pain relief method for acute, short-term pain in newborns.

A research protocol examining the effect of vibration on the crying duration variable in needle-related medical procedures in newborns also predicted that vibration therapy would be effective in reducing pain caused by vaccine injection and shortening the newborn's crying time.

The use of hands is the oldest known and universal method for relieving pain. Methods such as manual pressure application (similar to the flick method) are used to reduce pain during invasive procedures.

Manual methods can be incorporated into clinical practice without additional cost or time. Experimental and clinical studies have suggested that various types of manual stimulation of certain nerve fibers (manipulations such as rubbing, applying pressure, and tapping just above or below painful areas) followed by the release of beta-endorphin into the bloodstream relieves pain.

Flicking the injection site can be used to control pain in childhood. To date, only one experimental study testing the flick method has reported that the flick method applied before intramuscular injection had lower pain scores in babies during and after vaccination.

Studies show that the positive effects of both methods are mentioned. However, no study has been found to examine the effects of both methods on injection pain that may occur when the second dose of Hepatitis B vaccine is administered in the neonatal period and compare their effects. The fact that the effects of mechanical vibration and flicking methods as pain relief strategies on reducing pain, physiological parameters and crying duration have not been examined in this population before shows the deficiency in the literature. This study will be the first to examine the effectiveness of vibration analgesia with the flick method in intramuscular injection pain in the newborn baby population in the same sample group and to compare the analgesic effectiveness of both methods.

In line with all this information, this study aimed to examine the effect of flicking the injection site before the second dose of the Hepatitis B vaccine applied to the anterior surface of the vastus lateralis muscle in infancy and applying mechanical vibration to the injection site throughout the vaccination procedure on acute pain, crying duration and physiological parameters that may occur due to intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* Mothers agreeing to participate in the study,
* The baby's gestational age being between 38 and 42 weeks,
* Babies being 30-42 days old after birth,
* The baby's birth weight being between 2500 g and 4000 g
* The infant has not been given pain medication prior to vaccination and has a normal body temperature.

Exclusion Criteria:

* Araştırmaya katılmayı kabul etmeyen anneler,
* Gestasyonel yaşı 38. haftanın altında 42. haftanın üzerinde olan bebekler,
* Konjenital hastalık veya doğumsal anomalisi olan bebekler olarak belirlendi.

Ages: 30 Days to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Newborn infant pain assessment | The behavioral states of the infants were recorded with NIPS one minute before the procedure. The infants' responses to the pain they felt during the procedure were recorded with NIPS during the procedure. The infants' behavioral responses to pain after
  Before, during, and after the procedure, infants' behavioral responses to pain were recorded using NIPS.
body temperature measurement | Body temperature was measured one minute before the procedure. Body temperature was measured one minute after the procedure.
  Body temperature was measured before and after the procedure.
respiratory rate measurement | Respiratory rate was measured for 1 minute before the procedure began. Respiratory rate was measured until the first minute after the procedure.
  The infants' respiratory rate was measured before and after the procedure.
Oxygen saturation measured | Oxygen saturation was measured one minute before the procedure, during the procedure, and for one minute after the procedure.
  Oxygen saturation was measured before, during, and after the procedure.
heart rate measured | Heart rate was measured one minute before the procedure, during the procedure, and up to the first minute after the procedure.
  Heart rate was measured before, during, and after the procedure.
Crying duration measurement | With the start of the vaccination process, the crying duration was recorded on the Newborn Observation Form for one minute. The start of the procedure and the crying duration were recorded for one minute.
  The crying time was measured for one minute after the procedure.

SECONDARY OUTCOMES:
Newborn infant pain assessment | One minute before the procedure, behavioral responses to pain were recorded using NIPS. During the procedure, behavioral responses to pain were recorded using NIPS. Behavioral responses to pain were recorded using NIPS for one minute after the procedure.
  The infants' behavioral responses to pain were recorded before the procedure. During the procedure, the infants' behavioral responses to pain were recorded using NIPS. After the procedure, the infants' behavioral responses to pain were recorded using NIPS. Pain was rated on a scale of 0 (no pain) to 7 (highest level of pain).
Body temperature measured. | Body temperature was measured one minute before and one minute after the procedure.
  Body temperature was measured before and after the procedure.
Respiratory rate measured | Respiratory rate was measured for 1 minute before the procedure began. Respiratory rate was measured until the first minute after the procedure.
  The infants' respiratory rate was measured before and after the procedure.
oxygen saturation measured | Oxygen saturation was measured one minute before the procedure, during the procedure, and up to the first minute after the procedure.
  Oxygen saturation was measured before, during, and after the procedure.
Heart rate measured | Heart rate was measured one minute before the procedure, during the procedure, and for one minute after the procedure.
  Heart rate was measured before, during, and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: BERRİN GÖGER, LECTURER, Principal Investigator — GU, KSDHSV School, Department of Medical Services and Techniques, Gümüşhane, Türkiye
Locations (1):
- Kelkit No. 1 Family Health Center, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No. There are no plans to share individual participant data.

REFERENCES:
- See also: Principal investigator Berrin GÖGER's institutional affiliation web address — https://kelkitshmyo.gumushane.edu.tr/tr/
- See also: Principal investigator Berrin GÖGER's institutional affiliation web address — http://kelkitshmyo.gumushane.edu.tr/tr/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT07185152/Prot_SAP_000.pdf
  • Study Protocol and Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT07185152/Prot_ICF_001.pdf